CLINICAL TRIAL: NCT01002326
Title: An Open Trial of Cognitive-Behavioral Therapy (CBT) for Pediatric Body Dysmorphic Disorder (BDD)
Brief Title: Cognitive-Behavioral Therapy for Pediatric Body Dysmorphic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sabine Wilhelm, Director, OCD and Related Disorders Program at Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008P002270
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Body Dysmorphic Disorder
Keywords: Pediatric; Body Dysmorphic Disorder; BDD; CBT; Cognitive-Behavioral Therapy
MeSH Terms: conditions — Body Dysmorphic Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive-Behavioral Therapy (Experimental)
  Interventions: Behavioral: Cognitive-Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy — 20 sessions of Cognitive-Behavioral Therapy

SUMMARY:
The purpose of this study is to develop and test the effectiveness of Cognitive-Behavioral Therapy (CBT) for children and adolescents suffering from Body Dysmorphic Disorder.

DETAILED DESCRIPTION:
The main purpose of this trial is to develop and investigate the effects of a CBT protocol for children and adolescents with BDD. It is important to investigate CBT in this population given the disorder's early onset and poor trajectory if left untreated.

In the first phase of this trial, we will develop the treatment manual, adapting the adult manual for use in a pediatric population. In the second phase of this trial we will test the effectiveness of the CBT treatment in 12 pediatric BDD patients. We intend to treat 12 children and adolescents with BDD. All patients will receive CBT. We will also examine treatment feasibility and acceptability (e.g., retention and reasons for treatment refusal and dropout, expectancy, and motivation), and we will explore predictors of outcome. Therapeutic progress will be broadly assessed with measures of beliefs, behaviors, mood, functioning, and quality of life before, during, and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DSM-IV BDD or its delusional variant, which must be present currently and for at least 6 months prior to study entry
* Total score of at least 24 on the 12-item BDD-YBOCS, adolescent version, which includes a score of at least 2 on item 1 (1-3 hours/day of preoccupation with the perceived defect)
* Score of at least moderate on the Clinical Global Impressions of Severity (CGI-Severity)
* Score of < 60 on the Child Global Assessment Scale (C-GAS)
* Ability to communicate meaningfully with the investigators and competent to provide written assent; both parental informed consent and adolescent assent must be obtained

Exclusion Criteria:

* Alcohol or substance abuse or dependence within the past 3 months, bipolar disorder, psychosis, organic mental disorder, development disorder, body image concerns accounted for primarily by an eating disorder or weight concerns. If subjects have another comorbid diagnosis, the BDD has to be the primary concern.
* Recent (within the past 6 months) suicide attempt, or suicidal ideation as indicated by a K-SADS score of 4 or higher that is active or warrants consideration of hospitalization
* Need for inpatient or partial hospital treatment
* Current psychotherapy and failure to benefit from ten or more sessions of previous CBT treatment
* Participants can be receiving psychotropic medication, but they must be on a stable dose for 2 months prior to the study baseline assessment and maintain this dosage throughout the course of the study

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2009-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale Modified for BDD (BDD-YBOCS)-Pediatric Version | Baseline, Monthly, Post-Treatment, 3-Month Follow-Up, 6-Month Follow-Up

SECONDARY OUTCOMES:
Brown Assessment of Beliefs Scale (BABS)-Pediatric Version | Baseline, Monthly, Post-Treatment, 3-Month Follow-Up, 6-Month Follow-Up
Clinical Global Impression Scale (CGI) | Baseline, Monthly, Post-Treatment, 3-Month Follow-Up, 6-Month Follow-Up
Children's Depression Inventory (CDI) | Baseline, Weekly, Post-Treatment, 3-Month Follow-Up, 6-Month Follow-Up

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, Ph.D., Principal Investigator — Massachusetts General Hospital; Jennifer Greenberg, Psy.D., Study Director — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States